CLINICAL TRIAL: NCT02102438
Title: Neoadjuvant or Adjuvant Chemotherapy Without Anthracyclines for Elderly Patients Diagnosed With HER2 Positive Breast Cancer
Brief Title: Chemotherapy for Elderly Patients Diagnosed With Localized HER2 Positive Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No financial support aproved
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP 477
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer; HER-2 Positive Breast Cancer
Keywords: Elderly patients; Localized HER2+ Breast Cancer; Omission of anthracyclines; Neoadjuvant chemotherapy; Adjuvant chemotherapy; Safety information
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trastuzumab and weekly chemotherapy (Experimental): Treatment schedule Weekly paclitaxel and Carboplatin at 80mg/m2 and Area under the curve (AUC) of 2, respectively. Weekly trastuzumab will be combined with chemotherapy (at a loading dose of 4mg/kg and a maintenance dose of 2mg/kg). Chemotherapy will be given at D1, D8 and D15 in a 28-day cycle, for a total of 4 treatment cycles.
  After completion of four chemotherapy cycles, Trastuzumab will be given at a dose of 6mg/kg every 21 days, for a total 14 cycles.
  Interventions: Drug: Trastuzumab; Drug: Weekly Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab (at a loading dose of 4mg/kg and a maintenance dose of 2mg/kg) will be given concomitantly with chemotherapy.
  After completion of four chemotherapy cycles, Trastuzumab will be given at a dose of 6mg/kg every 21 days, for a total 14 cycles.
  Other Names: Other names; Herceptin
Drug: Weekly Paclitaxel — Weekly paclitaxel at 80mg/m2 at D1, D8 and D15 in a 28-day cycle, for a total of 4 treatment cycles.
  Other Names: Taxol
Drug: Carboplatin — Carboplatin at an Area Under the Curve (AUC) of 2 at D1, D8 and D15 in a 28-day cycle, for a total of 4 treatment cycles.
  Other Names: Other names; Paraplatin

SUMMARY:
There is major concern regarding chemotherapy related toxicity in the group of women older than 65 years old diagnosed with human epidermal growth factor receptor 2 (HER2) positive breast cancer (BC). Nevertheless, these patients are at a particularly high risk of breast cancer recurrence and death. Of note, older patients may experience higher risk for Trastuzumabe related cardiotoxicity, especially when this agent is combined with an anthracycline.

Recent studies have shown extremely favourable outcomes in early HER2+ BC patients treated with a combination of paclitaxel and trastuzumab, omitting anthracyclines from treatment.

Investigators sought to investigate safety and outcome data on a cohort of elderly patients treated with weekly paclitaxel combined with carboplatin and trastuzumab.

DETAILED DESCRIPTION:
Breast cancer is the most common female cancer and the second most common cause of cancer death in women. BC incidence is markedly increased with aging.

Amplification or overexpression of HER2 oncogene is present in approximately 18 to 20% of primary invasive BC. In the absence of HER2 target therapy combined with adjuvant or neoadjuvant chemotherapy, HER2 overexpression or amplification is associated with high rates of disease recurrence and death.

There is major concern regarding chemotherapy related toxicity in the group of women older than 65 years old diagnosed with HER2 positive breast cancer. Nevertheless, these patients are at a particularly high risk of breast cancer recurrence and death. Of note, older patients may experience higher risk for Trastuzumabe related cardiotoxicity, especially when this agent is combined with an anthracycline.

Recent studies have shown extremely favourable outcomes in early HER2+ BC patients treated with a combination of paclitaxel and trastuzumab, omitting anthracyclines from treatment.

Investigators sought to investigate safety and outcome data on a cohort of elderly patients treated with weekly paclitaxel combined with carboplatin and trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Clinical or Pathological Stage I- IIIA breast adenocarcinoma.
* HER2 overexpression or amplification defined by immunohistochemistry staining of +3 or positive fluorescence in situ hybridization (FISH) test.
* Age ≥ 65 years old.
* WHO performance status less than 2; adequate hematologic (granulocyte count ≥ 2 X 109/L, platelet count ≥100 X109/L) and hepatic (transaminases ≤ 1.5 X the upper limit of normal (ULN), alkaline phosphatases ≤ 2.5 times ULN, and bilirubin ≤ ULN) tests; and normal cardiac function (baseline left ventricular ejection fraction at least ≥ 55%)

Exclusion Criteria:

* Radiologic imaging of metastatic disease.
* History of cardiac disease contraindicating anthracyclines, uncontrolled essential hypertension or diabetes, stroke or any other comorbidity that could potentially compromise chemotherapy treatment, such as chronic obstructive pulmonary disease.
* Any previous treatment with anti HER2 therapy.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) | 3 years
  Disease Free Survival was defined as the time from randomization until first relapse (local, regional, or distant), contralateral breast cancer, or death from any cause.

SECONDARY OUTCOMES:
survival (OS) | 2 years
  Secondary end points are overall survival (OS), defined from the time from randomization until death from any cause, and safety.

CONTACTS AND LOCATIONS:
Overall Officials: Debora de Gagliato, MD, Principal Investigator — Instituto do Cancer do Estado de São Paulo; Max Se Mano, MD phD, Study Chair — Instituto do Cancer do Estado de São Paulo
Locations (1):
- ICESP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
no data avalilable